CLINICAL TRIAL: NCT05085353
Title: Fetal Outcomes Among Pregnant Emergency General Surgery Patients: a Prospective Multi-center Evaluation of Pregnant Patients Undergoing Emergency General Surgery
Brief Title: Fetal Outcomes Among Pregnant Emergency General Surgery Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 076.TRA.2019.D
Record Dates: First submitted 2021-10-07; First posted 2021-10-20 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Complications; Acute Appendicitis; Acute Cholecystitis; Biliary Pancreatitis; Bowel Obstruction; Acute Diverticulitis
MeSH Terms: conditions — Pregnancy Complications; Appendicitis; Cholecystitis, Acute; Intestinal Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: non-obstetric acute general surgical disease — non-obstetric acute general surgical disease

SUMMARY:
Approximately 1 in 500 pregnant women require non-obstetric surgery. Surgical care for the pregnant woman raises concern for complications adversely affecting pregnancy outcomes. The most common reason for surgery is acute appendicitis followed by gallbladder disease. Despite the common incidence of non-obstetric surgery among pregnant women, little is known regarding fetal outcome and the impact of laparoscopic interventions versus traditional open procedures. Even less is known about the role of non-operative management of general surgical disease in the pregnant population. However, fetal outcome is not compromised by emergency general surgery condition interventions.

DETAILED DESCRIPTION:
Approximately 1 in 500 pregnant women require non-obstetric surgery. Surgical care for the pregnant woman raises concern for complications adversely affecting pregnancy outcomes. The most common reason for surgery is acute appendicitis followed by gallbladder disease. Despite the common incidence of non-obstetric surgery among pregnant women, little is known regarding fetal outcome and the impact of laparoscopic interventions versus traditional open procedures. Even less is known about the role of non-operative management of general surgical disease in the pregnant population. However, fetal outcome is not compromised by emergency general surgery condition interventions. The primary objective of this study is to establish best practices for management of pregnant patients requiring emergency non-obstetric general surgery.

This is a prospective multi-center observational study of pregnant women and their fetus/neonate (birth to 30 days) with acute general non-obstetric surgical diseases, including those undergoing operative and non-operative management. Data collected will be purely observational and involve no study-based therapeutic interventions or alterations in patient care. The patients will be managed per institutional standard of care. Data collection will occur in the following format:

* Initiated upon admission for general surgery until discharge for that admission
* Upon the birth of the child
* Post-delivery of the child, through that admission until discharged, for a maximum of 30 days post- delivery All of the data will be collected from the medical record, as long as the subject's providers utilize EPIC. Otherwise, an approved member of the research team may need to contact the patient via telephone to obtain access to their non-EPIC record.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 or older with non-obstetric acute general surgical disease (Acute appendicitis, Acute cholecystitis, Acute biliary pancreatitis, Bowel obstruction, Acute diverticulitis

Exclusion Criteria:

* Trauma patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women 18 or older with non-obstetric acute general surgical disease
Study Population: pregnant women and their fetus/neonate (birth to 30 days) with acute general non-obstetric surgical diseases, including those undergoing operative and non-operative management.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
past medical history/comorbidities | birth to 30 days
  Baseline demographics
prenatal care prior to surgery | birth to 30 days
  Baseline demographics
medical care within one year of conception | birth to 30 days
  Baseline demographics
disease process | birth to 30 days
  Baseline demographics

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Burris, MD, Principal Investigator — Trauma Center at Methodist Dallas Medical Center
Locations (1):
- Trauma Center at Methodist Dallas Medical Center, Dallas, Texas, United States